CLINICAL TRIAL: NCT02430532
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of BG00012 in Delaying Disability Progression in Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: BG00012 and Delay of Disability Progression in Secondary Progressive Multiple Sclerosis
Acronym: INSPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 109MS308; 2014-003021-18 (EudraCT Number)
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis, Secondary Progressive
Keywords: INSPIRE; SPMS; Tecfidera; BG00012
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dimethyl fumarate (Experimental): BG00012 120 mg (1 BG00012 120 mg capsule + 1 matching placebo capsule) orally twice daily (BID) for 1 week, followed by BG00012 240 mg orally BID thereafter.
  Interventions: Drug: dimethyl fumarate; Other: Placebo
- Placebo (Experimental): BG00012 120 mg capsule orally once a day supplemented with matching placebo capsules for the first 4 weeks of treatment, as an additional blinding measure. Matched placebo capsules only thereafter.
  Interventions: Drug: dimethyl fumarate; Other: Placebo

INTERVENTIONS:
Drug: dimethyl fumarate — capsule
  Other Names: DMF; BG00012; Tecfidera
Other: Placebo — matched placebo capsule

SUMMARY:
The primary objective of the study is to investigate whether treatment with BG00012 (dimethyl fumarate) compared with placebo slows the accumulation of disability not related to relapses in participants with secondary progressive multiple sclerosis (SPMS). The secondary objective of the study is to assess the effect of BG00012 compared with placebo on patient-reported outcomes, brain atrophy, and cognitive function.

ELIGIBILITY:
Key Inclusion Criteria:

* Onset of SPMS at least 1 to 2 years prior to randomization. SPMS is defined as relapsing-remitting disease followed by progression of disability independent of or not explained by relapses.
* Have documented confirmed evidence of disease progression independent of clinical relapses over the 1 year prior to randomization.
* Have an Expanded Disability Status Scale score of 3.0 to 6.5, inclusive.
* Have a Multiple Sclerosis (MS) Severity Score of 4 or higher.

Key Exclusion Criteria:

* Have a diagnosis of relapsing remitting multiple sclerosis or primary progressive MS as defined by the revised McDonald criteria.
* Had a recent clinical relapse (within 3 months) prior to randomization.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; serious or acute liver, kidney, or bone marrow dysfunction; uncontrolled diabetes; serious or acute psychiatric illness that would limit compliance with study requirements.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- United States (7):
  - Research Site, Long Beach, California
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Charlotte, North Carolina
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Round Rock, Texas
- Research Site, Brussels, Belgium
- Czechia (2):
  - Research Site, Brno
  - Research Site, Hradec Králové
- Research Site, Sittard-Geleen, Netherlands
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Plewiska
  - Research Site, Poznan
- Research Site, Banská Bystrica, Slovakia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: BG00012 120 mg capsule orally once a day (QD) supplemented with matching placebo capsules for the first 4 weeks of treatment. Matched placebo capsules only thereafter for up to 108 weeks.
- Tecfidera 240 mg BID: BG00012 120 mg orally twice daily (BID) for 1 week, followed by BG00012 240 mg orally BID beginning on Day 8 for up to 108 weeks.
Period: Overall Study
Arm/Group | Placebo | Tecfidera 240 mg BID
Started | 30 | 28
Completed | 0 | 0
Not Completed | 30 | 28
Not completed — Sponsor Decision to Stop Study Early | 30 | 25
Not completed — Consent Withdrawn | 0 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: BG00012 120 mg capsule orally QD supplemented with matching placebo capsules for the first 4 weeks of treatment. Matched placebo capsules only thereafter for up to 108 weeks.
- Tecfidera 240 mg BID: BG00012 120 mg orally BID for 1 week, followed by BG00012 240 mg orally BID beginning on Day 8 for up to 108 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tecfidera 240 mg BID | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (6.67) | 49.6 (8.05) | 50.2 (7.33)
Age, Customized [Number; unit: participants]
  < 20 years | 0 | 0 | 0
  20 to 29 years | 0 | 0 | 0
  30 to 39 years | 1 | 4 | 5
  40 to 49 years | 10 | 8 | 18
  >= 50 years | 19 | 16 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Time to Disability Progression Independent of Relapse
Description: Time to onset of confirmed progression of disability is defined as 1 or more of the following criteria, confirmed at ≥ 6 months after start of treatment and at Week 108 using 1 or more of the following assessments: Expanded Disability Status Scale (EDSS) score increased from Baseline of ≥ 1 point if baseline EDSS ≤ 5.5, or ≥ 0.5 point if Baseline EDSS ≥ 6.0; Timed 25-Foot Walk (T25FW) ≥ 20% increase from Baseline in the time taken for the 25-foot walk; worsening on the 9-Hole Peg Test (9HPT; ≥ 20% increase from Baseline in the time taken for the 9HPT, confirmed in the same hand). The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. The T25FW is a quantitative mobility and leg function performance test where the participant is timed while walking for 25 feet. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs.
Time Frame: Up to 108 weeks
Population: The limited number of participants enrolled and the early termination of the study resulted in efficacy data not collected, and efficacy outcomes not analyzed, as per the pre-specified plan of analysis.
Arm/Group | Placebo | Tecfidera 240 mg BID
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline to 2 Years on the 12-Item Multiple Sclerosis Walking Scale (MSWS-12)
Description: MSWS-12 is a participant self-assessment of walking limitations due to multiple sclerosis (MS) during the past 2 weeks. It contains 12 items that measure the impact of MS on walking. Items are summed to generate a total score and transformed to a scale with a range of 0 to 100, where high scores indicate greater negative impact on walking.
Time Frame: Baseline, 2 years
Population: as for outcome 1
Arm/Group | Placebo | Tecfidera 240 mg BID
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline to Week 108 in ABILHAND Questionnaire Score
Description: The ABILHAND Questionnaire measures the participant's perceived difficulty in performing everyday manual activities in the last 3 months. Participants fill in the 56-item questionnaire by estimating their own difficulty or ease in performing each of the 56 activities. Items are summed to generate a total score and transformed to a scale with a range of 0 to 100, where high scores indicate greater impact on manual ability.
Time Frame: Baseline, Week 108
Population: as for outcome 1
Arm/Group | Placebo | Tecfidera 240 mg BID
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage Change From Baseline to Week 108 in Whole Brain Volume
Description: Whole brain volume is measured by magnetic resonance imaging (MRI).
Time Frame: Baseline, Week 108
Population: as for outcome 1
Arm/Group | Placebo | Tecfidera 240 mg BID
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline to Week 108 in Cognitive Function as Measured by the Symbol Digit Modalities Test (SDMT)
Description: The SDMT measures the time to pair abstract geometric symbols with specific numbers. The score is the number of correctly coded items from 0-110 in 90 seconds. A higher score indicates a better outcome.
Time Frame: Baseline, Week 108
Population: as for outcome 1
Arm/Group | Placebo | Tecfidera 240 mg BID
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 24 weeks (overall mean time on study of 14.34, with an overall mean time on study treatment of 9.58 weeks).
Description: Data summaries of adverse events are descriptive in nature and the comparison between treatment groups might not be appropriate due to the small number of participants and limited study follow-up duration.
Arm/Group | Placebo | Tecfidera 240 mg BID
Serious Adverse Events (participants affected / at risk) | 0/30 | 5/28
Other Adverse Events (participants affected / at risk) | 9/30 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Tecfidera 240 mg BID (N=28)
Enteritis (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Tecfidera 240 mg BID (N=28)
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 2
Multiple sclerosis relapse (Nervous system disorders) | 0 | 2
Flushing (Vascular disorders) | 5 | 5

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor for business reasons. Efficacy, patient-reported outcomes, and pharmacodynamic data were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.